CLINICAL TRIAL: NCT03026153
Title: Biologics Anchoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB00040495
Record Dates: First submitted 2017-01-13; First posted 2017-01-20 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Moderate-to-severe Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - Oral Survey 1 (Other): Oral survey 1 will be administered as control intervention: patients will be asked how willing they would be to take an injectable medication to control their psoriasis which required once-monthly injections
  Interventions: Behavioral: Control Group Oral Survey 1
- Intervention Group - Oral Survey 2 (Other): Oral Survey 2 will be administered as the intervention : patients will be asked how willing they would be to take an injectable medication to control their psoriasis which required once-daily injections, then surveyor would ask how willing they would be to take an injectable medication which required only once-monthly injections
  Interventions: Behavioral: Intervention Group Oral Survey 2

INTERVENTIONS:
Behavioral: Control Group Oral Survey 1 — Oral survey 1 will be administered as control intervention: patients will be asked how willing they would be to take an injectable medication to control their psoriasis which required once-monthly injections
  Arms: Control group - Oral Survey 1
Behavioral: Intervention Group Oral Survey 2 — Oral Survey 2 will be administered as the intervention: patients will be asked how willing they would be to take an injectable medication to control their psoriasis which required once-daily injections, then surveyor would ask how willing they would be to take an injectable medication which required only once-monthly injections
  Arms: Intervention Group - Oral Survey 2

SUMMARY:
Biologics are used to treat conditions such as moderate-to-severe psoriasis, a chronic condition that impairs quality of life as much or more than other major medical conditions. Biopharmaceuticals are medications which are are isolated from biological sources including microorganisms, animals or humans. These medications generally function to decrease inflammation or disrupt the inflammatory cycle. Patients are often apprehensive about choosing a biologic medication over other options due to anxiety regarding the need for regular injections, leaving the patient undertreated and continuing to suffer with psoriasis. Reducing fears of injections may improve adherence to treatment and may improve treatment outcomes. Fear of injection is inherently subjective and may be easily modified. Anchoring is the tendency for humans to rely on a specific value when making decisions and to make judgments relative to that value. Patients who have never taken an injection will subjectively view the idea of taking an injection relative to the "not taking any injection" baseline. This comparison is scary and represents a considerable hurdle to taking a new injectable medication that may be otherwise optimal for their treatment. Resetting the anchor may be all that is needed to help patients overcome fear of injection. The objective is to assess whether patients offered a once monthly injectable biologic would be more likely to accept that biologic medication if they are first counseled about a daily injection.

DETAILED DESCRIPTION:
Biologics are used to treat a variety of medical conditions across multiple medical specialties. In the Dermatology specialty, biologics are used to treat conditions such as moderate-to-severe psoriasis, a chronic condition that impairs quality of life as much or more than other major medical conditions. Biopharmaceuticals are medications which are are isolated from biological sources including microorganisms, animals or humans. Examples of biologic medications commonly used in dermatology include tumor necrosis factor-alpha (TNF-alpha) blockers/inhibitors (etanercept, infliximab, certolizumab pegol, golimumab), interleukin 12/23 blockers (ustekinumab), and interleukin 17A blockers (secukinumab, ixekizumab).

These medications generally function to decrease inflammation or disrupt the inflammatory cycle. Biologic medications are administered via injection by the patient or a healthcare provider. Most of the medications require periodic injections approximately once per month. Patients may undergo periodic lab monitoring to assess for side effects. Biologic medications have revolutionized dermatology and the general medical field. Patients are often apprehensive about choosing a biologic medication over other option due to anxiety regarding the need for regular injections, leaving the patient undertreated and continuing to suffer with psoriasis. Reducing fears of injections may improve adherence to treatment and may improve treatment outcomes. Fear of injection is inherently subjective and may be easily modified.

Anchoring is the tendency for humans to rely on a specific value when making decisions and to make judgments relative to that value. Patients who have never taken an injection will subjectively view the idea of taking an injection relative to the "not taking any injection" baseline. This comparison is scary and represents a considerable hurdle to taking a new injectable medication that may be otherwise optimal for their treatment.

Resetting the anchor may be all that is needed to help patients overcome fear of injection. The investigators hypothesize that if a patient were first counseled about the possibility of taking an injectable biologic medication daily, they would be much less hesitant to take a monthly injection.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe psoriasis
* not currently managed with biologic or other injectable medication

Exclusion Criteria:

* Individuals younger than 18 (line of questioning necessary for the study may be beyond understanding in this age group)
* Currently managed with biologic medication or other injectable medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03-16 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Oral survey responses Oral Survey Outcomes | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Feldman, MD,PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Dept of Dermatology, WFUHS, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandler D, Bewley A. Biologics in dermatology. Pharmaceuticals (Basel). 2013 Apr 17;6(4):557-78. doi: 10.3390/ph6040557. PMID 24276125
- [Background] Wilson TD, Houston CE, Etling KM, Brekke N. A new look at anchoring effects: basic anchoring and its antecedents. J Exp Psychol Gen. 1996 Dec;125(4):387-402. doi: 10.1037//0096-3445.125.4.387. PMID 8945789